CLINICAL TRIAL: NCT04793776
Title: Manage Emotions to Reduce Aggression - MERA: A Brief Aggression Treatment for Veterans With PTSD Symptoms
Brief Title: Manage Emotions to Reduce Aggression (MERA)
Acronym: MERA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency); University of South Florida (Other); VA Boston Healthcare System (U.S. Federal Agency); University of Houston (Other); Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MHBP-007-20S; CX002135 (Other Grant/Funding Number: VA Clinical Science Research & Development)
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Stress Disorders, Post-Traumatic; Aggression; Emotion Regulation
Keywords: Stress Disorders, Post-Traumatic; Aggression; Emotion Regulation; Veterans; Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Aggression; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial (RCT) is designed to examine if a brief emotion regulation treatment, MERA, is efficacious at reducing aggression compared to present centered therapy (PCT) in Veterans with full or subthreshold PTSD. The investigators will use a parallel group RCT design, a 1:1 allocation ratio, and a superiority (MERA > PCT) framework. The study will follow the SPIRIT 2013 Checklist that is recommended for RCT protocols.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and outcome assessors will be masked to treatment assessment. Therapist will be masked to outcome data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manage Emotions to Reduce Aggression (MERA) (Experimental): MERA is 3 individual 90-minute sessions delivered over 3 weeks.
  Interventions: Behavioral: Manage Emotions to Reduce Aggression
- Present Centered Psychotherapy (PCT) (Active Comparator): PCT delivered in 3 individual 90-minute sessions over 3 weeks.
  Interventions: Behavioral: Present Centered Psychotherapy

INTERVENTIONS:
Behavioral: Manage Emotions to Reduce Aggression — MERA begins with education about the adaptive nature of emotions, how childhood and military experiences can influence emotion regulation, and how combat requires different emotion regulation strategies than most civilian environments. MERA use modeling and practice with feedback to teach cognitive-behavioral and acceptance-based emotion regulation skills.
  Other Names: MERA
  Arms: Manage Emotions to Reduce Aggression (MERA)
Behavioral: Present Centered Psychotherapy — PCT will serve as the comparison group. PCT assists Veterans in understanding and coping with current difficulties, such as aggression, but does not provide systematic training in emotion regulation skills.
  Other Names: PCT
  Arms: Present Centered Psychotherapy (PCT)

SUMMARY:
PTSD is one of the most prevalent mental health conditions affecting Veterans who have served since 9/11. Veterans with posttraumatic stress disorder (PTSD) report difficulty controlling impulsive aggression (IA). An inability to manage one's emotions (emotion dysregulation) is an underlying mechanism of IA. Reducing IA and increasing use of PTSD evidence-based psychotherapies are two critical missions for the Veterans Health Administration. The proposed research supports these missions by comparing a 3- session emotion regulation treatment (Manage Emotions to Reduce Aggression) to a control group in order to determine if MERA can reduce IA and prepare Veterans for PTSD treatment. By enhancing Veterans' abilities to cope with trauma-related emotions and feel equipped to initiate PTSD treatments, this research aims to help Veterans decrease IA and ultimately recover from PTSD.

DETAILED DESCRIPTION:
Aggression can have devastating interpersonal and societal consequences, including incarceration, family violence, disruption of treatment-facilitating factors, and death. About 50% of Veterans with full and subthreshold posttraumatic stress disorder (PTSD) reported engaging in aggression after returning from deployment. This level of aggression is higher than Veterans without PTSD5 and civilians with PTSD. Current psychotherapy options to reduce aggression include present centered therapies (PCTs), anger management, and evidence based psychotherapies (EBP) for PTSD. Anger management reduces aggression in civilian samples with small to moderate effect sizes. However, few anger management treatment studies have examined Veterans with PTSD and measured acts of aggression. Consistently, VA clinicians also provide PCTs and EBP for PTSD. It is unknown how effectively PCTs reduce aggression. Unfortunately, even with gold standard EBP for PTSD Veterans only experience small to moderate reductions in aggression. While any decline is an improvement, these treatments leave room for novel methods to help Veterans reduce aggression.

Emotion regulation ability may be a key to reducing aggression. The team revealed that among Veterans with PTSD and aggression, impulsive aggression (emotionally charged, reactive, and uncontrolled) is more common than premeditated aggression (deliberate, instrumental, and planned). Emotion dysregulation, or the inability to detect emotions, accept emotions, and/or engage in content-appropriate regulation, is related to impulsive aggression and to PTSD severity. The investigators demonstrated that emotion dysregulation fully mediated the relationship between PTSD and impulsive aggression in Veterans.

Increasing emotion regulation ability of many emotions is an innovative method to reduce aggression. Full-length treatments that incorporate emotion regulation training (8-12 sessions) have augmented EBP for PTSD and improved Veterans' emotion regulation skills. However, a brief format is needed for returning Veterans. Eight weeks of treatment, particularly when offered prior to EBP, is an unfeasible commitment for many Veterans who are reintegrating into their communities. Additionally, most drop outs from EBP for PTSD occur prior to session three making the initial sessions a critical time for skill development. Finally, Veterans have experienced wait times to receive treatment due to the growing population of returning Veterans. To address these challenges, the team developed a 3-session emotion regulation treatment, called Manage Emotions to Reduce Aggression (MERA). Male combat Veterans who completed MERA in an open trial (N=20) endorsed the brief model, utilized the skills, and found the treatment helpful at the 4-week follow up. MERA had a low dropout rate of 8% from active treatment. MERA completers demonstrated a medium to large pre- to post-treatment reduction in frequency of aggression (Cohen's d = 0.73).

The goal of the proposed study is to conduct a 2-site randomized clinical trial (RCT) to test if MERA is efficacious at reducing aggression and emotion dysregulation compared to 3 sessions of PCT, which is often the standard of care for Veterans with aggression.

Aim 1: Determine if MERA results in reductions in frequency of impulsive aggression compared to PCT in Veterans (N = 204) with subthreshold or full PTSD who have deployed for combat operations since 9/11.

Hypothesis 1: MERA will demonstrate statistically significant greater reductions in frequency of aggression (measured by the Overt Aggression Scale) relative to PCT at the 2-month posttreatment assessment.

Aim 2: Examine if MERA reduces emotion dysregulation relative to PCT. Hypothesis 2: MERA will demonstrate statistically significant greater reductions in emotion dysregulation (measured by Difficulties in Emotion Regulation Scale) relative to PCT at the posttreatment assessment.

Exploratory Aim. Veterans who learn to regulate their emotions rather than avoid them may be more likely to engage in EBP for PTSD. The investigators will examine if Veterans who complete MERA have higher rates of EBP initiation compared to Veterans who complete PCT. Exploratory Hypothesis: Veterans who complete MERA will have statistically significant higher rates of EBP initiation than Veterans who complete PCT.

If the hypotheses are supported, the VA will have a brief treatment that can help Veterans manage their aggression by directly targeting emotion dysregulation. MERA may also be applicable to Veterans with emotion dysregulation and other psychological disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female Veterans who deployed to combat zones since 9/11.
2. Currently meets criteria for full or subthreshold PTSD, determined by the Clinician-Administered PTSD Scale for DSM-5
3. Engaged in at least 3 self-reported aggressive acts (e.g., yelling, throwing objects, hitting objects/people) in the last month, measured by the Overt Aggression Scale
4. Impulsive aggression is his/her primary form of aggression, determined by the Impulsive Premeditated Aggression Scale
5. Each Veteran must allow an independent aggression rater (live-in partner, family member, or roommate above 18 years of age)] verify the number of aggressive acts, using the Overt Aggression Scale.
6. Agreement not to change psychotropic medications through the duration of the study.

Exclusion Criteria:

1. Currently suicidal with intent of self-harm in the last week.
2. Currently homicidal with plans to hurt a specific person.
3. Unable to complete self-report measures.
4. Meets diagnostic criteria for bipolar disorder or psychotic disorder.
5. Had a psychotropic medication change within 4 weeks prior to the baseline assessment. Veterans receiving general mental health services or engaging in usual care will be allowed to participate.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Overt Aggression Scale (OAS) | Treatment group differences in change from Session 1 to posttreatment assessment (duration of 11 weeks).
  Overt Aggression Scale is a 17-item self-report measure that assesses frequency of verbal and physical aggression against self, other, and objects and while driving over the past week. Veterans' self-reported aggressive acts will be summed to create an OAA total score. Minimum score = 0; there is no maximum score as Veterans can report as many episodes of aggression as they engage in.

SECONDARY OUTCOMES:
Change in Difficulties in Emotion Regulation Scale (DERS) | Treatment group differences in change from Session 1 to posttreatment assessment (duration of 11 weeks).
  Difficulties in Emotion Regulation Scale (16) is a 36-item self-report measure with 6 different emotion-dysregulation factors: nonacceptance of emotional responses, difficulties engaging in goal directed behaviors, impulse-control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. Scoring is based on how well the item describes the individual in the past month, from 1 (almost never) to 5 (almost always). Minimum score = 36; Maximum score = 180. Higher scores represent more emotion dysregulation.

OTHER OUTCOMES:
Evidence Based Psychotherapy (EBP) Initiation | Treatment group differences in EBP initiation at 6 months posttreatment.
  Initiation is defined as attending at least 1 Prolonged Exposure, Cognitive Processing Therapy, or Eye Movement Desensitization and Reprocessing session. EBP for PTSD initiation is assessed at 6 months posttreatment via chart review. Scores can either be 0 = Did not begin EBP or 1 = began EBP.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon R. Miles, PhD, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (2):
- United States (2):
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying publications resulting from the proposed research will be shared outside VA in electronic format through the mechanism(s) indicated below.
  * A De-identified, Anonymized Dataset will be created and shared.
  * Final de-identified data sets underlying publications resulting from the proposed research will be available outside the VA using the following mechanism, electronic format through e-mail upon request, after results are published. Data sets will also be available through collaborators and other investigators upon request prior to publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After results of study are published.
Access Criteria: After results of study are published and according to the VA record control schedule, which is currently a maximum of 6 years.